CLINICAL TRIAL: NCT02616965
Title: A Phase I Trial Assessing the Feasibility of Romidepsin Combined With Brentuximab Vedotin for Patients Requiring Systemic Therapy for Cutaneous T-cell Lymphoma
Brief Title: A Study to Assess the Feasibility of Romidepsin Combined With Brentuximab Vedotin in Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Seagen Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-085; 16-1009 (Other: Fox Chase cancer Center)
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous T-cell Lymphoma (CTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — romidepsin; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment consists of the combination of Romidepsin given 10mg/m2 or 14mg/m2 on days 1, 8 and 15 every 28 days and Brentuximab vedotin given 0.9mg/kg or 1.2mg/kg on days 1 and 15 every 28 days for 16 cycles.
  Interventions: Drug: Romidepsin; Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Romidepsin — Romidepsin at the dosage 10mg/m2 or 14mg/m2 will be given ONCE 14 days prior to cycle one and then on days 1,8,15 in each cycle. Each cycle is 28 days and treatment will continue up to 16 cycles
Drug: Brentuximab vedotin — Brentuximab vedotin at the dosage 0.9mg/kg or 1.2 mg/kg will be given on days 1 and 15 in each cycle. Each cycle is 28 days and treatment will continue up to 16 cycles

SUMMARY:
This is a Phase I Trial to assess the feasibility of Romidepsin combined with Brentuximab Vedotin for patients requiring Systemic Therapy for Cutaneous T-cell Lymphoma.

DETAILED DESCRIPTION:
This is a traditional "3+3" phase 1 dose de-escalation design testing up to 3 dose levels of romidepsin in conjunction with brentuximab vedotin in patients with untreated or previously treated (up to 2 prior systemic regimens, including photopheresis) CTCL. Dose-limiting toxicities (DLT) will be determined during cycle 1. The first 3 subjects will begin at dose level 1. If no DLT is encountered another 3 subjects will be enrolled at the same dose level. The maximum tolerated dose (MTD) will be the dose level at which ≤ 1 of 6 of subjects experience DLT. If more than one subject at any one dose level encounters a DLT, the dose will be de-escalated for all subsequent subjects. Should no DLTs occur, the investigators will not escalate beyond dose level 1. Once the MTD has been confirmed, the investigators will enroll an additional 9 patients in a toxicity refinement cohort for a total of 15 evaluable patients at the MTD.

Treatment will continue for up to 16 cycles (one cycle is 28 days) or until disease progression or toxicities, whichever occurs first. Drugs can be continued after 16 cycles if a patient has derived a clinical benefit from treatment after discussion with the sponsor-investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed diagnosis of mycosis fungoides (MF), Sezary syndrome (SS) or primary cutaneous CD30-positive lymphoproliferative disorder, including lymphomatoid papulosis and primary cutaneous ALCL (pc-ALCL)as defined by the WHO classification of Tumors of Hematopoietic and Lymphoid tissue.

   Please note that tumor samples for patients with MF or SS can be CD30 negative and do not have to be CD30 positive on either flow cytometry or immunohistochemistry for patients to be eligible.
2. Patients with MF/SS must have stage IB, IIA, IIB, III or IV disease; patients with primary cutaneous CD30-positive lymphoproliferative disorder must have multifocal symptomatic or extensive lesions requiring systemic treatment.
3. Patients must require systemic treatment.
4. Patients can have received up to 2 lines of systemic treatment. Psoralen plus ultraviolet light therapy (PUVA) is not considered to be a systemic therapy.
5. Age > 18 years.
6. ECOG performance status 0, 1 or 2.
7. Patients must have acceptable organ and marrow function as defined below:

   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Total bilirubin within normal institutional limits
   * AST/ALT (SGOT/SGPT) < 2 times institutional normal limits
   * Creatinine within normal institutional limits OR
   * Creatinine clearance > 60 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal
8. Women of child-bearing potential (WOCBP) must have a negative pregnancy test
9. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
10. Patients with HIV who are not receiving cytochrome p450 inhibitors, and who have a minimum of 300+ CD4+ cells/mm3, an undetectable viral load, and no history of AIDS indicator conditions.

Exclusion Criteria:

1. Patients who have not had resolution of clinically significant toxic effects of prior anticancer therapy to ≤grade 1 as per by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI-CTCAE, v.4.0).
2. Grade 2 or greater neuropathy.
3. Patients may not be receiving any other investigational agents.
4. Patients with known CNS involvement.
5. Patients must not receive concurrent systemic or topical steroids or other skin directed therapy while on study except as outlined in 5.2.2
6. Patients who have experienced allergic reactions to monoclonal antibodies.
7. Patients who have received prior HDAC inhibitors, or brentuximab vedotin, except for patients who were exposed to above drugs only for a short time (less than 8 weeks), did not progress while on treatment, and did not have intolerable toxicity but were discontinued for another reason (e.g., comorbidity) may be permitted to enter the study after discussion with the sponsor-investigator.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant or breast feeding. Refer to section 4.4 for further detail.
10. Second malignancies that require active treatment with the exception of breast or prostate cancer on endocrine therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | during treatment period which is an average of 64 weeks.
  CTCAE v4.03
Dose-limiting toxicities (DLTs) | during the first 28 days (cycle 1) of treatment
  CTCAE v4.03

SECONDARY OUTCOMES:
overall safety and tolerability of the combination of brentuximab vedotin & romidepsin assessed by adverse events. | from start of treatment to 30 days post treatment period (16 cycles)
  CTCAE v4.03
Estimate complete and partial response rate of the combination treatment | 64 weeks, 30 days post treatment and every 12 weeks post-treatment, up to 2 years
  mSWAT skin assessment
Estimate complete and partial response rate of the combination treatment | 64 weeks, 30 days post treatment and every 12 weeks post-treatment, up to 2 years
  Global Response Score (GRS).
Overall survival (OS) | From the time of patient registration until death, measured every 12 weeks up to 2 years
  OS is measured by length of time
Progression free survival (PFS) | From the time of patient registration until disease progression, measured every 12 weeks up to 2 years
  PFS is measured in length of time by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Nakhoda, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - University of Pennsylvania, Perelman Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No